CLINICAL TRIAL: NCT02053584
Title: Dario™ Blood Glucose Monitoring System - User Performance Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LabStyle Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR-0002
Record Dates: First submitted 2014-01-30; First posted 2014-02-03 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2016-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dario BGMS (Experimental)
  Interventions: Device: Dario™ Blood Glucose Meter; Device: YSI2003

INTERVENTIONS:
Device: Dario™ Blood Glucose Meter — Each subject will undergo a finger prick and also provide a venous blood sample
Device: YSI2003 — Blood samples will be tested using YSI (gold standard) for comparison to evaluate accuracy.

SUMMARY:
The study is performed to evaluate the accuracy of blood glucose level results obtained from fingertip using Labstyle Dario Blood Glucose Monitoring System (BGMS) compared to reference equipment (YSI 2300 STATPLUS) and to evaluate the ease of use of the Dario Device by the lay-person.

The participants will review the Dario user manual and guide and will be requested to operate the Dario BGMS and perform their own glucose blood test, after which they will be asked to complete a questionnaire. As reference the participants will be tested by professional caregivers both using the Dario BGMS and by YSI 2003.

DETAILED DESCRIPTION:
Device accuracy will be assessed based on the acceptance criteria of ISO 15197:2003 which states: "The minimum acceptable accuracy for results produced by a glucose monitoring system shall be as follows: 95% of the individual glucose results shall fall within 15 mg/dL of the results of Reference method at glucose concentrations ≥ 4,2 mmol/L (≥ 75 mg/dL)".

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the age 18 and 80
* Type 1 and Type 2 diabetes

Exclusion Criteria:

* Drug and alcohol abuse
* Investigator discretion

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2013-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Vainstein, MD, Principal Investigator — Wolfson Medical Center

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 230 patients were consented, the patients from day one (n=68) were excluded from the final results analysis due to a number of technical issues.
Period: Overall Study
Arm/Group | Dario BGMS
Started | 230
Completed | 230 (68 subjects (day one participants) were excluded from the final analysis.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dario BGMS
Number analyzed (Participants) | 161
Age, Continuous [Median (Standard Deviation); unit: years] | 55.5 (17.6)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 95
  >=65 years | 66
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 64
Region of Enrollment [Number; unit: participants]
  Israel | 161

OUTCOME MEASURES:

1. Primary Outcome: BGMS Accuracy Assessment When Used by Layperson
Description: The minimum acceptable accuracy for results produced by a glucose monitoring system shall be as follows: 95% of the individual glucose results shall fall within 15 mg/dL of the results of reference method (YSI) at glucose concentrations ≥ 4,2 mmol/L (≥ 75 mg/dL). (ISO 15197:2003)
Time Frame: Within 6 seconds of applying blood drop to strip
Measure: Number; unit: percentage of participants
Arm/Group | Dario BGMS
Number analyzed (Participants) | 161
percentage of participants
  < 75 mg/dl Within ±5mg/dL | 2
  < 75 mg/dl Within ±10mg/dL | 4
  < 75 mg/dl Within ±15mg/dL | 6
  >= 75 mg/dl Within ±5% | 44
  >= 75 mg/dl Within ±10% | 78
  >= 75 mg/dl Within ±15% | 126
  >= 75 mg/dl Within ±20% | 150
  >= 75 mg/dl | 155

2. Secondary Outcome: Evaluation of the Ease of Use of the Dario BGMS by the Lay-person
Description: Each participant receives a survey to fill in describing their usage of the device and their opinions on the ease of use.
Time Frame: Within a couple of hours from the time labelling material was provided to the subject
Measure: Number; unit: participants
Groups:
- Dario BGMS (Easily Understood): Dario™ Blood Glucose Meter: Each subject will undergo a finger prick and also provide a venous blood sample. Subjects reported that the labels were easily understood.
  YSI2003: Blood samples will be tested using YSI (gold standard) for comparison to evaluate accuracy.
- Dario BGMS (Understood After Few Attempts): Dario™ Blood Glucose Meter: Each subject will undergo a finger prick and also provide a venous blood sample. Subjects reported that the labels were understood after few attempts.
  YSI2003: Blood samples will be tested using YSI (gold standard) for comparison to evaluate accuracy.
- Dario BGMS (Did Not Understand How to Use): Dario™ Blood Glucose Meter: Each subject will undergo a finger prick and also provide a venous blood sample. Subjects reported that the labels were not clear and that they did not understand how to use.
  YSI2003: Blood samples will be tested using YSI (gold standard) for comparison to evaluate accuracy.
Arm/Group | Dario BGMS (Easily Understood) | Dario BGMS (Understood After Few Attempts) | Dario BGMS (Did Not Understand How to Use)
Number analyzed (Participants) | 161 | 161 | 161
participants | 93 | 67 | 1

ADVERSE EVENTS:
Arm/Group | Dario BGMS
Serious Adverse Events (participants affected / at risk) | 0/161
Other Adverse Events (participants affected / at risk) | 0/161

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No